CLINICAL TRIAL: NCT07095959
Title: Marshall Vein Ethanol Infusion in Addition to Pulsed Electric Field Ablation Versus Pulsed Electric Field Ablation Alone for Paroxysmal Atrial Fibrillation
Acronym: MARVEL-PAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Caihua Sang, Executive director of Arrhythmia center, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MARVEL-PAF
Record Dates: First submitted 2025-07-22; First posted 2025-07-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFA-PVI + EIVOM group (Experimental): PVI will be performed with PFA first, then EIVOM will be performed to achieve potential cardiac autonomous nerve modulation while reinforce LPV isolation.
  Interventions: Procedure: vein of Marshall ethanol infusion; Procedure: PVI using pulsed field ablation
- PFA-PVI group (Active Comparator): PVI will be performed with PFA only
  Interventions: Procedure: PVI using pulsed field ablation

INTERVENTIONS:
Procedure: vein of Marshall ethanol infusion — After PFA, the coronary sinus venography will be acquired in search of VOM ostium. Then an over-the-wire balloon will be sent into the VOM and deflated with 4-6 atm. Selective VOM venography will be performed, followed by injection of 10ml 95% ethanol into the VOM.
  Arms: PFA-PVI + EIVOM group
Procedure: PVI using pulsed field ablation — Bilateral pulmonary vein antrum ablation using a pulsed field ablation

SUMMARY:
The Marvel-PAF trial is an investigator initiated, multi-center, open-label, randomized trial, which aims to compare the effectiveness of vein of Marshall in addition to pulmonary vein isolation using pulsed field ablation in the treatment of paroxysmal atrial fibrillation. The primary endpoint is any atrial arrhythmias lasting ≥30s without AAD during 12 months after procedure excluding the 2-months blanking period.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years;
2. With symptomatic* paroxysmal AF;
3. Undergoing first AF ablation;
4. At least one AF lasting over 30s documented by 12-lead ECG, Holter, or other rhythm monitoring device in the past 12 months;
5. Able to understand the purpose of the study, willing to receive randomization of the ablation strategy, and able to be followed up as required, voluntarily participate in the study and signed a written informed consent.

   * Symptoms include but not restricted to palpitations, dizziness, fatigue, or shortness of breath and chest discomfort

Exclusion Criteria:

1. Diagnosed with persistent atrial fibrillation or duration of atrial fibrillation >7 days;
2. Thrombosis in the heart cavity;
3. Contraindications to oral anticoagulants including the presence of a history of heparin-induced thrombocytopenia;
4. Transient/reversible atrial fibrillation due to electrolyte disorders, thyroid disease or other non-cardiac-related causes;
5. Acute coronary syndrome in the past 3 months or coronary intervention or coronary artery bypass treatment;
6. Stroke or transient ischemic attacks (TIA) in the past 3 months;
7. History of cardiac surgery or other surgical history involving left atrium, such as previous left atrial catheter ablation, atrial septal defect repair, etc.;
8. History of previous severe valvular disease (severe mitral stenosis or regurgitation), congenital heart disease, hypertrophic cardiomyopathy or dilated cardiomyopathy;
9. TEE examination in the past 12 months showed that the left atrium diameter of the parasternal long axis section was ≥55mm;
10. Other factors that are not suitable for surgery (such as history of organ transplant surgery or ongoing evaluation of organ transplant surgery, life expectancy less than 1 year, uncontrolled cancer, pregnancy, breastfeeding, or planning to get pregnant, etc.);
11. Other patients who were not suitable for enrollment in this study after the investigator's evaluation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Any atrial arrhythmias lasting ≥30s without AAD during 12 months after procedure excluding the 2-months blanking period | 12 months after procedure excluding the 2-month blanking period

SECONDARY OUTCOMES:
Any atrial arrhythmias lasting ≥30s with or without AAD during 12 months after procedure excluding the 2-months blanking period | 12 months after procedure excluding the 2-months blanking period
Any atrial flutter/atrial tachycardia lasting ≥30s during 12 months after procedure excluding the 2-months blanking period | 12 months after procedure excluding the 2-months blanking period
Any atrial arrhythmias after multiple ablation with or without AADs | 12 months after first procedure excluding the 2-months blanking period
AF burden | 12 months after procedure excluding the 2-months blanking period
  Total AF/AFL time devided by total monitoring time
procedural complications | 30 days after the procedure
Change in quality of life | at baseline and 12 months after procedure
  Assessed by AFEQT scale

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual data will be shared only upon reasonable request to the principal investigator